CLINICAL TRIAL: NCT00152646
Title: Platelets Induced Vasodilation, in Vitro and in Vivo Study in Patients With Arteriopathy and Healthy Subjects.
Brief Title: Platelets Induced Vasodilation, in Vitro and in Vivo Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PHRC 04-07
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Last update posted 2010-02-04 (Estimated); Status verified 2005-09

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: placebo, aspirine, clopidogrel

SUMMARY:
The aim of the study is to show the implication of platelets in vasodilation using in vivo and in vitro analysis and to compare the effects of placebo, aspirin and Clopidogrel in this interaction platelets/vessels.

The effects of 7 days of each treatment will be compared in healthy subjects and patients with arteriopathy.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria healthy subjects

* Man or Woman 18 years
* Agreement signed
* French health insurance
* Able to understand the study
* Biological haemostatic test normal
* Vascular Doppler of lower limbs normal
* Pressure index > 1 in both lower limbs

Inclusion criteria healthy subjects

* Man or Woman 18 years
* Agreement signed
* French health insurance
* Able to understand the study
* Biological haemostatic test normal
* Lower limbs arteriopathy (clinical, pressure index, Doppler)

Exclusion Criteria:

* Unable to sign agreement
* Subjects protected by low
* Participation to other study
* Changes of treatment within the 15 days before inclusion
* Chronic treatment with Clopidogrel or drugs against inflammation
* Severe respiratory, cardiac, kidney, hepatic insufficiency
* Haemostatic troubles
* Diabetic neuropathy
* Neurologic desease (Parkinson…..)
* Hypertension
* Symptomatic stomach ulcer
* Anaemia Hb<11g/l
* Pregnant women or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2005-03; Study Completion 2008-01 (Estimated)

PRIMARY OUTCOMES:
In vivo vasodilation induced by low intensity current
In vitro study of platelets function
In vitro vasodilation induced by platelets in isolated rat's vessels

CONTACTS AND LOCATIONS:
Overall Officials: Marc Antoine Custaud, MD PhD, Principal Investigator — University Hospital, Angers
Locations (1):
- Exploration Fonctionnelles Vasculaires, Angers, Maine et Loire, France